CLINICAL TRIAL: NCT04351230
Title: Phase II Trial of Abemaciclib and T-DM1 in Women and Men With HER2-positive Advanced or Metastatic Breast Cancer Who Progressed on Treatment With a Taxane, Trastuzumab and Pertuzumab
Brief Title: T-DM1 With or Without Abemaciclib for the Treatment of HER2-Positive Metastatic Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: There are no patients enrolled on this study and all efforts are being discontinued
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACCRU-BR-1801; NCI-2020-02218 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCRU-BR-1801 (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2020-04-15; First posted 2020-04-17 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-02

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; HER2 Positive Breast Carcinoma; Metastatic Breast Carcinoma; Prognostic Stage IV Breast Cancer AJCC v8
MeSH Terms: conditions — Breast Neoplasms | interventions — abemaciclib; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (trastuzumab emtansine) (Active Comparator): Patients receive trastuzumab emtansine IV over 90 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Trastuzumab Emtansine
- Arm B (trastuzumab emtansine, abemaciclib) (Experimental): Patients receive trastuzumab emtansine IV over 90 minutes on day 1 and abemaciclib PO BID on days 1-21. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Abemaciclib; Biological: Trastuzumab Emtansine

INTERVENTIONS:
Drug: Abemaciclib — Given IV
  Other Names: LY-2835219; LY2835219; Verzenio
  Arms: Arm B (trastuzumab emtansine, abemaciclib)
Biological: Trastuzumab Emtansine — Given PO
  Other Names: Ado Trastuzumab Emtansine; ADO-Trastuzumab Emtansine; Kadcyla; PRO132365; RO5304020; T-DM1; Trastuzumab-DM1; Trastuzumab-MCC-DM1; Trastuzumab-MCC-DM1 Antibody-Drug Conjugate; Trastuzumab-MCC-DM1 Immunoconjugate

SUMMARY:
This phase II trial studies how well T-DMI with or without abemaciclib works for the treatment of HER2-positive breast cancer that has spread to other places in the body (metastatic). T-DM1 is a monoclonal antibody, called trastuzumab, linked to a chemotherapy drug called DM1. Trastuzumab attaches to HER2 positive cancer cells in a targeted way and delivers DM1 to kill them. Abemaciclib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving T-DM1 and abemaciclib may work better in treating patients with breast cancer compared to T-DM1 alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess whether progression-free survival (PFS) is improved with the addition of abemaciclib to trastuzumab emtansine (T-DM1) for patients with estrogen receptor positive (ER+)HER2-positive advanced or metastatic breast cancer who progressed on treatment with a taxane, trastuzumab and pertuzumab (Cohort 1).

II. To assess whether progression-free survival (PFS) is improved with the addition of abemaciclib to T-DM1 for patients with estrogen receptor negative (ER-) HER2-positive advanced or metastatic breast cancer who progressed on treatment with a taxane, trastuzumab and pertuzumab (Cohort 2).

SECONDARY OBJECTIVES:

I. To assess the safety and tolerability of each treatment regimen. II. To assess overall survival (OS) and objective response rate (ORR) of each treatment regimen.

CORRELATIVE RESEARCH OBJECTIVES:

I. To assess whether the presence of vimentin expression or the level of tumor infiltrating lymphocytes (TILs) in the baseline tumor specimen is associated with an increased likelihood of longer PFS in the abemaciclib arms compared to the non-abemaciclib arms (regardless of ER status).

II. To assess both the baseline prognostic effects of circulating tumor cell (CTC) levels, ER expression in CTCs, HER2 expression in CTCs, serum TK1 levels, circulating tumor-derived deoxyribonucleic acid (ctDNA), ESR1, or PIK3CA mutations and whether a reduction in these levels after 2 cycles of treatment is associated with an increased likelihood of longer PFS overall and separately in the treatment arms.

III. To assess whether polymorphisms in FCgamma receptors (FCGR2A and FCGR3A) are associated with inferior PFS.

IV. To describe alterations seen in the peripheral blood immune system architecture after 2 cycles of treatment.

V. To assess whether peripheral blood immune markers at baseline are prognostic and whether change in peripheral blood immune markers after 2 cycles of treatment are associated with PFS.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive T-DM1 intravenously (IV) over 90 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive T-DM1 IV over 90 minutes on day 1 and abemaciclib orally (PO) twice daily (BID) on days 1-21. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION - INCLUSION CRITERIA
* Agree to undergo a core biopsy of breast cancer tissue derived from a local, regional or distant site for mandatory confirmation of ER+/ER-, progesterone receptor (PR) and HER2 status

  * NOTE: If a single lesion is present, imaging must be completed after the lesion is biopsied and measurements must be taken from this image for disease evaluation by Response Evaluation Criteria in Solid Tumors (RECIST) to be considered eligible for this trial
  * NOTE: The study requires a fresh biopsy for clinical and research purposes and archival tissue does not suffice. If the patient has already undergone a biopsy at the time of disease progression prior to enrolling on the trial, an additional research biopsy will still be required
* Imaging or histologic evidence of progression of unresectable locally advanced or metastatic breast cancer
* One of the following must be true:

  * Progressed/relapsed during or within 12 months of completing neo-adjuvant treatment with a regimen containing a taxane, trastuzumab and pertuzumab
  * Progressed/relapsed during or within 12 months of completing adjuvant treatment with a regimen containing a taxane, trastuzumab and pertuzumab
  * Progressed/relapsed during metastatic treatment with a regimen containing a taxane, trastuzumab and pertuzumab
  * Progressed/relapsed > 12 months after receipt of adjuvant T-DM1
* A total of 1 or 2 prior lines of the following breast cancer therapies in any disease setting

  * Chemotherapy alone
  * HER2-directed therapy alone
  * Chemotherapy with HER2 directed therapy
  * Note: Any number of prior lines of endocrine therapy received in any disease setting
* Measurable disease as defined by RECIST criteria

  * NOTE: Tumor lesions in a previously irradiated area are not considered measurable disease. Disease that is measurable by physical examination only is not eligible
* Eastern Cooperative Oncology Group (ECOG) performance status (PS): 0 or 1
* Left ventricular ejection fraction (LVEF) >= 50% as determined by echocardiography or multiple-gated acquisition imaging =< 21 days prior to pre-registration
* Able to swallow oral medication
* Provide written informed consent =< 28 days prior to pre-registration
* Willingness to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Willingness to provide mandatory tissue specimens for correlative research
* RANDOMIZATION - INCLUSION CRITERIA
* Local, histological confirmation of metastatic HER2-positive breast cancer per American Society of Clinical Oncology (ASCO) College of American Pathologists (CAP) guidelines; one of the following must apply

  * 3+ by immunohistochemistry (IHC)
  * 2+ by IHC and in situ hybridization (ISH) amplified
* Discontinued all cancer therapies (chemotherapy, radiotherapy, immunotherapy, and endocrine therapy), except trastuzumab, >= 21 days prior to randomization for myelosuppressive agents or >= 14 days prior to randomization for non-myelosuppressive agents

  * NOTE: All residual toxicities (except alopecia) should be at baseline or grade 1 (including peripheral neuropathy)
  * NOTE: If indicated, patients can commence treatment with bisphosphonates of RANK-L inhibitors (e.g., denosumab) any time prior to randomization. No washout period or treatment delay is required prior to commencing study treatment
* Absolute neutrophil count >= 1.5 x 10^9/L (obtained =< 14 days prior to randomization)
* Platelet count >= 100,000/mm^3 (obtained =< 14 days prior to randomization)
* Hemoglobin >= 9.0 g/dL (obtained =< 14 days prior to randomization)
* Creatinine =< 1.5 X upper limit of normal (ULN) (obtained =< 14 days prior to randomization)
* Total bilirubin =< 1.5 x ULN (obtained =< 14 days prior to randomization) (except in cases of known Gilbert's syndrome where =< 2.0 x ULN is allowed and direct bilirubin within normal levels is permitted)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN (obtained =< 14 days prior to randomization)

  * NOTE: If liver metastases are present, AST and ALT =< 5 x ULN are acceptable
* Prothrombin time (PT)/international normalized ratio (INR)/partial thromboplastin time (PTT) =< 1.5 X ULN OR if patient is receiving anticoagulant therapy and PT or PTT is within therapeutic range of intended use of coagulants (obtained =< 14 days prior to randomization)
* Negative pregnancy test =< 7 days prior to randomization, for persons of childbearing potential only

  * NOTE: A female of childbearing potential must have a negative serum pregnancy test within 7 days of the first dose of T-DM1 +/- abemaciclib and agree to use a highly effective contraception method during the treatment period and for 6 months following the last dose of T-DM1 +/- abemaciclib
  * Women and men of reproductive potential should agree to use an appropriate method of birth control throughout their participation in this study due to the teratogenic potential of the therapy utilized in this trial. Appropriate methods of birth control include abstinence, oral contraceptives, implantable hormonal contraceptives or double barrier method (diaphragm plus condom). Birth control must be used during the treatment period and continued for at least 6 months after the last dose of treatment with T-DM1 +/- abemaciclib
  * Cases of pregnancy that occur during maternal exposures to T-DM1+/- abemaciclib, or cases of pregnancy in female partners/spouses of male patients, should be reported. If a female patient is determined to be pregnant following T-DM1 +/- abemaciclib initiation, she must discontinue treatment immediately. Data on fetal outcome and breast-feeding are to be collected for regulatory reporting and drug safety evaluation
* Willingness to provide mandatory blood specimens for correlative research

Exclusion Criteria:

* PRE-REGISTRATION - EXCLUSION CRITERIA
* Any of the following prior therapies:

  * Surgery =< 21 days prior to pre-registration
  * Chemotherapy =< 21 days prior to pre-registration
  * Radiation =< 14 days prior to pre-registration
  * NOTE: Single fraction radiotherapy is allowed/exempt from this washout period
  * NOTE: Must have fully recovered from the toxicities of therapy, except for alopecia or peripheral neuropathy
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens

  * NOTE: Examples include interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline grade 2 or higher diarrhea
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy which interacts with the study drug(s)
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Or psychiatric illness/social situations that would limit compliance with study requirements
* Any of the following =< 14 days prior to pre-registration:

  * Active bacterial infection (requiring intravenous [IV] antibiotics)
  * Fungal infection,
  * Detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C)
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Other active non-breast malignancy =< 3 years prior to pre-registrations

  * EXCEPTIONS: Patients with a history of adequately treated cancers that are of very low risk of recurrence (i.e. papillary thyroid cancer treated with surgery, carcinoma in situ of the cervix, non-melanoma skin cancer) are eligible
  * NOTE: If there is a history of prior malignancy, the patient must not be receiving other specific anti-neoplastic treatment
* History of any of the following conditions:

  * Syncope of cardiovascular etiology
  * Ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation)
  * Sudden cardiac arrest
* History of myocardial infarction =< 6 months prior to pre-registration or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Received prior treatment with any CDK 4 and CDK 6 inhibitor (e.g. abemaciclib, ribociclib or palbociclib) or participated in any CDK 4 and CDK 6 inhibitor clinical trial for which treatment assignment is still blinded
* Received live virus vaccine =< 28 days prior to pre-registration
* Currently taking and unable to discontinue medications that are moderate or strong inhibitors and/or inducers of CYP3A or CYP3A4 before pre-registration
* Unstable or newly diagnosed brain metastases requiring local treatment

  * NOTE: Stable treated brain metastases allowed

    * Specifically, central nervous system metastasis are allowed provided they have been treated (i.e., surgery, radiation, and/or radiosurgery) >= 12 weeks prior to pre-registration and have stable neurologic function, including no requirement for medication(s) to control symptoms for >= 2 weeks prior to pre-registration
  * NOTE: Patients with known leptomeningeal disease are not eligible
* RANDOMIZATION - EXCLUSION CRITERIA
* Unable to provide histological confirmation of metastatic or locally advanced HER2-positive breast cancer per ASCO CAP guidelines
* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential who are unwilling to employ adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | The time elapsed between treatment initiation and tumor progression or death from any cause, assessed up to 5 years
  For each treatment arm, the distribution of PFS times will be estimated using the Kaplan-Meier method. A stratified log rank test) will be used to assess whether the PFS is increased with the addition of abemaciclib to trastuzumab emtansine (T-DM1). Also, a point and interval estimate of the hazard of progression with abemaciclib plus T-DM1 relative to the hazard of progression with abemaciclib alone with be obtained from the results of fitting a stratified Cox model with treatment arm as the covariate.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 5 years
  Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be used to grade and assign attribution to each adverse event reported. For each treatment arm, the proportion of patients who report developing a grade 2-5 of this adverse event (AE) will be determined.
Overall response rate (ORR) | Up to 5 years
  ORR is defined as the number of patients whose disease meets the Response Evaluation Criteria in Solid Tumors (RECIST) for a partial (PR) or complete (CR) on two consecutive evaluations at least 12 weeks apart divided by the total number of patients in that cohort who started protocol treatment. For each treatment arm, a 90% binomial confidence interval will be constructed for the true overall response rate.
Duration of response | Up to 5 years
  For the patients whose disease responded to treatment by meeting the criteria for CR or PR on two consecutive evaluations at least 12 weeks apart, the duration of response will be tabulated.
Overall survival (OS) | From randomization to death due to any cause, assessed up to 5 years
  Overall survival estimates for each treatment arm will be determined using the Kaplan Meier method. This study was not designed to compare the OS distributions of these 2 treatment regimens. As such, no hypothesis testing will be performed. A point and interval estimate of the hazard of death with abemaciclib plus T-DM1 relative to the hazard of progression with abemaciclib alone with be obtained from the results of fitting a stratified Cox model with treatment arm as the covariate.

CONTACTS AND LOCATIONS:
Overall Officials: Ciara C O'Sullivan, Principal Investigator — Academic and Community Cancer Research United
Locations (6):
- United States (6):
  - Yuma Regional Medical Center, Yuma, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Carle Cancer Center NCI Community Oncology Research Program, Urbana, Illinois
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin